CLINICAL TRIAL: NCT06791863
Title: Visceral Fat Area as a Prognostic Biomarker in Clear Cell Renal Cell Carcinoma: A Multicenter Study on Postoperative Survival
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 0361-02
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: ccRCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: The group with high area of body compositions (skeletal muscle, subcutaneous fat, subcutaneous fat or total fat)
- Cohort 2: the group with low area of body compositions (skeletal muscle, subcutaneous fat, subcutaneous fat or total fat)

SUMMARY:
This retrospective study included 1030 patients with clear cell renal cell carcinoma (ccRCC) who underwent radical or partial nephrectomy at Wuhan Union Hospital from 2014 to 2023.

ELIGIBILITY:
Inclusion Criteria:

1. primary clear cell renal cell carcinoma confirmed by histopathology;
2. patients≥18 years;
3. availability of preoperative abdominal computed tomography (CT) data;
4. patients with partial or radical nephrectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with clear cell renal cell carcinoma (ccRCC) who underwent radical or partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China